CLINICAL TRIAL: NCT03487705
Title: Clinical and Electrophysiological Characterization of Essential Tremor in Children and Adolescents
Brief Title: Essential Tremor in Children and Adolescent
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Halted Prematurely due to difficulties in inclusion.
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UF9770
Record Dates: First submitted 2018-02-01; First posted 2018-04-04 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-09

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- child essential tremor (Other): electromyogram with accelerometer
  Interventions: Other: electromyographic essential tremor

INTERVENTIONS:
Other: electromyographic essential tremor — * Making a recording electromyographic recording of the essential tremors in each child included at prospective.
  * Collect an electromyographic recording of essential tremors already made in each child included at retrospective.

SUMMARY:
Essential tremor (TE) is the most common abnormal movement of the adult. His diagnosis is based on a bundle of clinical arguments (Movement Disorders Society, 1998). Well characterized in the adult, little data is available concerning child. The objective of this work is (1) to define the demographic and clinical characteristics of the TE of children and adolescents, (2) to determine the electrophysiological characteristics in the child, (3) evaluate the functional impact of TE, and assess the functional impact of TE, and assess the current management modalities of TE in children and adolescent.

DETAILED DESCRIPTION:
A multicenter, descriptive cross-sectional study will include children and adolescents whose diagnosis of TE has been retained by an abnormal movement specialist before the age of 18 years.

Each child will benefit from an examination and a neurological and general clinical examination, a functional questionnaire, an electromyogram with accelerometer.

Will be determined: demographic characteristics (age, sex and ethnicity), family history of essential tremor, age of onset of tremor, tremor characteristics (location, occurrence conditions, aggravating or precipitating factors, scalability); additional examinations carried out and the treatments proposed or taken by the child as well as the functional repercussions of TE in the child.

Patients with tremor who meet the inclusion and exclusion criteria will be selected retrospectively or prospectively from the active queue of patients at each center.

ELIGIBILITY:
Inclusion Criteria:

* Subject whose age is between 3 and 18 years
* Subject affiliated to a social security scheme
* Parents or subjects who have been informed of the course and consequences of the study by an investigator and who have signed the informed consent form for prospective inclusion or who have given their non-opposition for retrospective inclusion.
* Diagnosis of essential tremor established according to the diagnostic criteria of the Movement Disorders Society (1998), by a neuropediatrician or a neurologist, specialist in abnormal movements. The diagnosis is based on the presence of the following criteria: bilateral action tremor of the hands and forearms, absence of other neurological signs.
* Availability of an electromyogram for retrospective inclusions.

Exclusion Criteria:

* Abnormal neurological examination outside tremor
* Family history or personal dysthyroidism
* Existence of a global psychomotor or motor developmental delay
* Taking medication that may induce tremor
* known poisoning by heavy metals, bismuth, mercury, methyl bromide
* Severe appearance of the tremor
* Tremor suggestive of a psychogenic origin
* Abnormal or non-existent brain MRI if family case

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
characteristics of TE | 1 day
  échelle Fahn-Marin- Tolosa FMT

SECONDARY OUTCOMES:
determine the electrophysiological characteristics impact of TE functional questionnaire, an electromyogram with accelerometer. | 1 day
  electromyogram with accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Agathe ROUBERTIE, Pr, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU Gui de Chauliac, Montpellier, France

IPD SHARING:
Plan to Share IPD: No